CLINICAL TRIAL: NCT00741689
Title: A Randomised, Single-Blind, Placebo-Controlled, Single-Centre, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single Ascending Oral Doses of AZD1656 in Japanese Healthy Male Volunteers
Brief Title: A Study to Evaluate Safety and Tolerability After Single Oral Dosing of AZD1656 in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: D1020C00003
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Volunteers
Keywords: Japanese; healthy; volunteers
MeSH Terms: interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- 1 (Experimental): AZD1656 in 6 increasing oral single doses given to 6 groups (5 on active and 1 on placebo in each group)
  Interventions: Drug: AZD1656

INTERVENTIONS:
Drug: AZD1656 — Dose escalation of oral single doses of AZD1656 to achieve maximal tolerated dose

SUMMARY:
The purpose of this study is to assess safety and tolerability of AZD1656 after single ascending oral doses in Japanese healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese males aged ≥20 and ≤40 years of age
* Clinically normal physical findings and laboratory values as judged by the investigator including negative test of Hepatitis B surface antigen, antibodies to HIV virus and antibodies to Hepatitis C virus

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within two weeks before the first administration of the IP
* History of psychiatric or somatic disease/condition that may interfere with the objectives of the study, as judged by the investigator.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety variables (AEs, blood pressure (BP), pulse, safety laboratory variables and electrocardiography (ECG) | Safety variables taken repeatedly during 24 hours on study day sessions

SECONDARY OUTCOMES:
Pharmacokinetic variables | Pharmacokinetic variables taken repeatedly during 24 hours on study day sessions
Pharmacodynamic variables | Blood samples taken repeatedly during 24 hours on study day sessions

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD Prof, Study Director — AstraZeneca R&D Mölndal; Mark Yen, MD, Principal Investigator — California Clinical Trials
Locations (1):
- Research Site, Glendale, California, United States

REFERENCES:
- [Derived] Ericsson H, Roshammar D, Wollbratt M, Heijer M, Persson M, Ueda S, Leonsson-Zachrisson M, Norjavaara E. Tolerability, pharmacokinetics, and pharmacodynamics of the glucokinase activator AZD1656, after single ascending doses in healthy subjects during euglycemic clamp. Int J Clin Pharmacol Ther. 2012 Nov;50(11):765-77. doi: 10.5414/CP201747. PMID 22943931